CLINICAL TRIAL: NCT02996474
Title: Pembrolizumab and Decitabine for Refractory or Relapsed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 170026; 17-H-0026
Record Dates: First submitted 2016-12-16; First posted 2016-12-19 (Estimated); Results first posted 2020-05-21 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2019-11-20

CONDITIONS: Relapsed Acute Myeloid Leukemia
Keywords: Pembrolizumab; Decitabine; AML (Acute Myelogenous Leukemia)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — pembrolizumab; Decitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab and Decitabine for treatment of Acute Myeloid Leukemia (Experimental): Pembrolizumab 200 mg will be administered as a 30 minute IV infusion every 3 weeks. Up to eight cycles of pembrolizumab will be given during the initial induction phase. Each cycle is 21 days. Decitabine will be administered at a dose of 20 mg/m^2 by intravenous infusion over approximately 1 hour repeated daily ordinarily on days 8 through 12 and 15 through 19 of alternative cycles (ie: cycles 1, 3, 5, 7) for treatment relapsed/refractory AML.
  Interventions: Drug: Pembrolizumab; Drug: Decitabine

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg will be administered as a 30 minute IV infusion every 3 weeks. Every effort should be made to target infusion timing to be as close to 30 minutes as possible. However, given the variability of infusion pumps, a window of -5 minutes and +10 minutes is permitted (i.e., infusion time is 30 minutes: -5 min/+10 min).
  Other Names: Keytruda; MK-3475
Drug: Decitabine — Will be administered at a dose of 20 mg/m^2 by continuous intravenous infusion over 1 hour repeated daily ordinarily on days 8 through 12 and 15 through 19 of alternative cycles (ie: cycles 1, 3, 5, 7). Decitabine should be repeated every 6 weeks.
  Other Names: Dacogen

SUMMARY:
Background:

Acute myeloid leukemia (AML) is a cancer of the white blood cells. It is fatal if not treated. Treatment for AML that has not responded to treatment (refractory) or has returned after treatment (relapsed) often do not work. Researchers want to see if an immunotherapy drug, combined with a less intense chemotherapy, may be able to help.

Objective:

To test if pembrolizumab, in combination with decitabine, is a possible treatment for people with relapsed or refractory AML.

Eligibility:

Adults 18 years of age and older with refractory AML or relapsed AML.

Design:

Participants will be first screened for eligibility.

The study is counted in 21-day cycles. The initial phase of the study consists of 8 cycles. Participants may be in the study for up to 2 years if they are responding to the treatment.

The first 3 weeks of treatment is usually done in the hospital. The rest may be done as an outpatient.

Participants will get pembrolizumab at the beginning of each cycle through an IV.

Participants will usually get decitabine by IV on days 8 12 and days 15 19 of every other cycle.

Participants will give blood samples.

Participants will have bone marrow exams. A needle will be inserted into the hip to extract cells from the bone marrow.

Some participants may give a sample of saliva from the inside of their cheek.

Some participants may give a small skin sample. The top layer of the skin is removed.

Some patients may require leukapheresis before starting treatment. This is a procedure to remove leukemia cells in the blood stream.

DETAILED DESCRIPTION:
This is a pilot study to determine the feasibility of a novel combination of Pembrolizumab and Decitabine in relapsed/refractory adult AML patients. While both Pembrolizumab and Decitabine are FDA approved agents, this study will explore giving these drugs in combination for this population of patients.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Unequivocal diagnosis of relapsed or refractory acute myeloid leukemia (AML) confirmed by an NIH attending pathologist within 30 days of study enrollment (includes residual AML as confirmed by institutional standards by NIH pathologists
* Received at least one prior AML therapy before study enrollment.
* Ability to comprehend the investigational nature of the study and provide informed consent.
* Be at least 18 years of age on day of signing informed consent.
* Availability of a physician willing to assume clinical care after completion of the study.
* Be willing to provide blood and bone marrow for research as described in the study.
* Have a performance status of less than or equal to 1 on the ECOG Performance Scale
* Demonstrate adequate organ function as defined below, all screening labs should be performed within 14 days of treatment initiation.
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential must be willing to use an adequate method of contraception; Contraception, for the course of the study through 120 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Male subjects of childbearing potential must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Adequate Organ Function Laboratory Values: System Laboratory - Value

  * Renal

    ---Serum Creatinine - Less than or equal to 1.5 X upper limit of normal (ULN)
  * Hepatic

    * Serum total bilirubin Less than or equal to 1.5 X ULN OR
    * Direct bilirubin less than or equal to ULN for subjects with total bilirubin levels greater than 1.5 ULN
    * AST (SGOT) and ALT(SGPT) Less than or equal to 3 X ULN

EXCLUSION CRITERIA:

The subject must be excluded from participating in the trial if the subject:

* Has a diagnosis of acute promyelocytic leukemia (APL)
* Has previously received an allogeneic hematopoietic stem cell transplant.
* Has received AML treatment with an investigational therapy or device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis)
* Has hypersensitivity to pembrolizumab or any of its excipients.
* Has hypersensitivity to decitabine or any of its excipients.
* Has received more than two prior cycles of decitabine.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1.

  --Note: Subjects who have received cytoreductive therapy with hydroxyurea at any time prior to study Day 1 are an exception to this criterion.
* Has not recovered (i.e., less than or equal to Grade 1 or at baseline) from adverse events due to previously administered AML therapy agents.

  * Note: Subjects with less than or equal to Grade 2 neuropathy are an exception and may qualify for the study.
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Patients with basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer would not be excluded.
* Has known malignant central nervous system (CNS) involvement.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has history of (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Has an active infection requiring intravenous systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject s participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist ) are live attenuated vaccines, and are not allowed.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-12-16; Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher S Hourigan, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Goswami M, Gui G, Dillon LW, Lindblad KE, Thompson J, Valdez J, Kim DY, Ghannam JY, Oetjen KA, Destefano CB, Smith DM, Tekleab H, Li Y, Dagur P, Hughes T, Marte JL, Del Rivero J, Klubo-Gwiezdzinksa J, Gulley JL, Calvo KR, Lai C, Hourigan CS. Pembrolizumab and decitabine for refractory or relapsed acute myeloid leukemia. J Immunother Cancer. 2022 Jan;10(1):e003392. doi: 10.1136/jitc-2021-003392. PMID 35017151
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-H-0026.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab and Decitabine for Treatment of Acute Myeloid Leukemia: Pembrolizumab 200 mg will be administered as a 30 minute IV infusion every 3 weeks. Up to eight cycles of pembrolizumab will be given during the initial induction phase. Each cycle is 21 days. Decitabine will be administered at a dose of 20 mg/m^2 by intravenous infusion over approximately 1 hour repeated daily ordinarily on days 8 through 12 and 15 through 19 of alternative cycles (ie: cycles 1, 3, 5, 7) for treatment relapsed/refractory Acute Myeloid Leukemia (AML).
Period: Overall Study
Arm/Group | Pembrolizumab and Decitabine for Treatment of Acute Myeloid Leukemia
Started | 10
Completed | 5
Not Completed | 5
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab and Decitabine for Treatment of Acute Myeloid Leukemia
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of a Novel Combination of Pembrolizumab and Decitabine in Relapsed/Refractory Acute Myeloid Leukemia Participants
Description: The number of patients who could be treated with a novel combination of Pembrolizumab and Decitabine in relapsed/refractory Acute Myeloid Leukemia participants without being removed from the protocol due to treatment related toxicities.
Time Frame: 24 weeks
Population: All patients enrolled on study.
Measure: Number; unit: Participants
Arm/Group | Pembrolizumab and Decitabine for Treatment of Acute Myeloid Leukemia
Number analyzed (Participants) | 10
Participants | 10

2. Secondary Outcome: Median Days to First Response From Start of Study to Initial Achievement of First Response (mCR, mCRi, CR, CRi, PR, or SD)
Description: Time to first response (days) is time from start of study to first response (mCR, mCRi, CR, CRi, PR, or SD) in relapsed/refractory acute myeloid leukemia (AML) participants.
  Measurable residual disease (MRD) negative complete remission is no evidence of residual disease, < 5% blasts, no Auer rods and may be with mCR or without count recovery (ANC ≥ 1,000/mcl and platelet count ≥ 100,000/mcl) as mCRi. Morphologic complete remission (CR) is ANC ≥ 1,000/mcl, platelet count ≥ 100,000/mcl, < 5% blasts, no Auer rods, no evidence of disease; Morphologic complete remission with incomplete blood count recovery (CRi) is same as CR but ANC may be < 1,000/mcl and/or platelet count < 100,000/mcl; Partial remission (PR) is ANC ≥ 1,000/mcl, platelet count > 100,000/mcl, and at least a 50% decrease in the percentage of marrow aspirate blasts to 5-25%, or marrow blasts < 5% with persistent Auer rods. Stable disease (SD) is absence of a complete or partial response, and no progressive disease.
Time Frame: At the end of each cycle 2 (week 6), 4 (week 12), 6 (week 18), 8 (up to week 24)
Population: Includes all participants that received treatment.
Measure: Median (Full Range); unit: days
Arm/Group | Pembrolizumab and Decitabine for Treatment of Acute Myeloid Leukemia
Number analyzed (Participants) | 10
days | 42 [37 to 49]

3. Secondary Outcome: Median Days to Best Response From Start of Study to Initial Achievement of Best Response (by the Order of mCR, mCRi, CR, CRi, PR, or SD)
Description: Time to Best Response is defined as time (days) from start of study to initial achievement of best response. Best response is defined by the order of mCR, mCRi, CR, CRi, PR, or SD. Measurable residual disease (MRD) negative complete remission is no evidence of residual disease, < 5% blasts, no Auer rods and may be with mCR or without count recovery (ANC ≥ 1,000/mcl and platelet count ≥ 100,000/mcl) as mCRi. Morphologic complete remission (CR) is ANC ≥ 1,000/mcl, platelet count ≥ 100,000/mcl, < 5% blasts, no Auer rods, no evidence of disease; Morphologic complete remission with incomplete blood count recovery (CRi) is same as CR but ANC may be < 1,000/mcl and/or platelet count < 100,000/mcl; Partial remission (PR) is ANC ≥ 1,000/mcl, platelet count > 100,000/mcl, and at least a 50% decrease in the percentage of marrow aspirate blasts to 5-25%, or marrow blasts < 5% with persistent Auer rods. Stable disease (SD) is absence of a complete or partial response, and no progressive disease.
Time Frame: At the end of each cycle 2 (week 6), 4 (week 12), 6 (week 18), 8 (up to week 24)
Population: Includes all participants that received treatment.
Measure: Median (Full Range); unit: days
Arm/Group | Pembrolizumab and Decitabine for Treatment of Acute Myeloid Leukemia
Number analyzed (Participants) | 10
days | 42 [39 to 159]

4. Secondary Outcome: Median Duration (Days) of Response From Initial Achievement of Response to Loss of Response (mCR, mCRi, CR, CRi, PR, or SD)
Description: To determine duration (days) of response as defined as time from initial achievement of response to loss of response (mCR, mCRi, CR, CRi, PR, or SD).
  Measurable residual disease (MRD) negative complete remission is no evidence of residual disease, < 5% blasts, no Auer rods and may be with mCR or without count recovery (ANC ≥ 1,000/mcl and platelet count ≥ 100,000/mcl) as mCRi. Morphologic complete remission (CR) is ANC ≥ 1,000/mcl, platelet count ≥ 100,000/mcl, < 5% blasts, no Auer rods, no evidence of disease; Morphologic complete remission with incomplete blood count recovery (CRi) is same as CR but ANC may be < 1,000/mcl and/or platelet count < 100,000/mcl; Partial remission (PR) is ANC ≥ 1,000/mcl, platelet count > 100,000/mcl, and at least a 50% decrease in the percentage of marrow aspirate blasts to 5-25%, or marrow blasts < 5% with persistent Auer rods. Stable disease (SD) is absence of a complete or partial response, and no progressive disease.
Time Frame: At the end of each cycle 2 (week 6), 4 (week 12), 6 (week 18), 8 (up to week 24)
Population: Includes all participants that received treatment.
Measure: Median (Full Range); unit: days
Arm/Group | Pembrolizumab and Decitabine for Treatment of Acute Myeloid Leukemia
Number analyzed (Participants) | 10
days | 148 [12 to 337]

5. Secondary Outcome: Median Duration (Days) of Best Response From Initial Achievement of Best Response to Loss of Best Response (by the Order of mCR, mCRi, CR, CRi, PR, or SD)
Description: Duration of Best Response is time (days) from initial achievement of best response to loss of best response. Best response is defined by the order of mCR, mCRi, CR, CRi, PR, or SD. Measurable residual disease (MRD) negative complete remission is no evidence of residual disease, < 5% blasts, no Auer rods and may be with mCR or without count recovery (ANC ≥ 1,000/mcl and platelet count ≥ 100,000/mcl) as mCRi. Morphologic complete remission (CR) is ANC ≥ 1,000/mcl, platelet count ≥ 100,000/mcl, < 5% blasts, no Auer rods, no evidence of disease; Morphologic complete remission with incomplete blood count recovery (CRi) is same as CR but ANC may be < 1,000/mcl and/or platelet count < 100,000/mcl; Partial remission (PR) is ANC ≥ 1,000/mcl, platelet count > 100,000/mcl, and at least a 50% decrease in the percentage of marrow aspirate blasts to 5-25%, or marrow blasts < 5% with persistent Auer rods. Stable disease (SD) is absence of a complete or partial response, and no progressive disease.
Time Frame: At the end of each cycle 2 (week 6), 4 (week 12), 6 (week 18), 8 (up to week 24)
Population: Includes all participants that received treatment.
Measure: Median (Full Range); unit: days
Arm/Group | Pembrolizumab and Decitabine for Treatment of Acute Myeloid Leukemia
Number analyzed (Participants) | 10
days | 148 [12 to 316]

6. Secondary Outcome: Overall Survival
Description: Number of participants overall survival is defined as death from any cause
Time Frame: from enrollment until date of death, assessed up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab and Decitabine for Treatment of Acute Myeloid Leukemia
Number analyzed (Participants) | 10
Participants | 0

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: The Adverse Event reporting period for this study begins when the patient takes the first dose of study drug and ends with the safety follow-up visit. If an Serious Adverse Event is present at the safety follow-up visit or within 30 days of the last dose of study drug (whichever is later), it should be followed to resolution or until the Investigator assesses the subject as stable, a new anticancer therapy is initiated, or the subject is lost to follow-up or withdraws consent.
Groups:
- Pembrolizumab and Decitabine for Treatment of Acute Myeloid Leukemia: Pembrolizumab 200 mg will be administered as a 30 minute IV infusion every 3 weeks. Up to eight cycles of pembrolizumab will be given during the initial induction phase. Each cycle is 21 days. Decitabine will be administered at a dose of 20 mg/m2 by intravenous infusion over approximately 1 hour repeated daily ordinarily on days 8 through 12 and 15 through 19 of alternative cycles (ie: cycles 1, 3, 5, 7) for treatment relapsed/refractory AML.
Arm/Group | Pembrolizumab and Decitabine for Treatment of Acute Myeloid Leukemia
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 7/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab and Decitabine for Treatment of Acute Myeloid Leukemia (N=10)
Febrile neutropenia (Blood and lymphatic system disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 1
Pain (General disorders) | 2
Sepsis (Infections and infestations) | 2
Wound infection bacterial (Infections and infestations) | 1
Blood culture positive (Investigations) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab and Decitabine for Treatment of Acute Myeloid Leukemia (N=10)
Increased tendency to bruise (Blood and lymphatic system disorders) | 3
Petechiae (Blood and lymphatic system disorders) | 4
Atrial flutter (Cardiac disorders) | 1
Cardiomegaly (Cardiac disorders) | 2
Dizziness (Cardiac disorders) | 2
Dyspnoea (Cardiac disorders) | 5
Localised oedema (Cardiac disorders) | 4
Oedema peripheral (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 3
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Diabetes insipidus (Endocrine disorders) | 1
Hyperglycaemia (Endocrine disorders) | 5
Hypoglycaemia (Endocrine disorders) | 2
Hypothyroidism (Endocrine disorders) | 2
Thyroid mass (Endocrine disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Eye pain (Eye disorders) | 2
Eye symptom (Eye disorders) | 1
Myopia (Eye disorders) | 1
Nystagmus (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Anorectal discomfort (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 2
Fecal incontinence (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 1
Lip ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Oral hemorrhage (Gastrointestinal disorders) | 1
Oral mucosal blistering (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 4
Perirectal abscess (Gastrointestinal disorders) | 1
Throat irritation (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Chills (General disorders) | 2
Decreased appetite (General disorders) | 4
Fatigue (General disorders) | 8
Gait disturbance (General disorders) | 1
Generalised oedema (General disorders) | 1
Head discomfort (General disorders) | 1
Hematoma (General disorders) | 1
Lethargy (General disorders) | 4
Malaise (General disorders) | 4
Non-cardiac chest pain (General disorders) | 3
Pain (General disorders) | 4
Pain in extremity (General disorders) | 1
Vascular access complication (General disorders) | 1
Vessel puncture site bruise (General disorders) | 1
Hepatomegaly (Hepatobiliary disorders) | 1
Hypoalbuminaemia (Hepatobiliary disorders) | 5
Enterococcal infection (Infections and infestations) | 1
Infections and infestations- Other, specify- Bacteremia (Infections and infestations) | 1
Paronychia (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Blister (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 2
Fracture (Injury, poisoning and procedural complications) | 2
Post-operative hemorrhage (Injury, poisoning and procedural complications) | 1
Skin wound (Injury, poisoning and procedural complications) | 1
Tendonitis (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 6
Alanine aminotransferase increased (Investigations) | 7
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 5
Blood alkaline phosphatase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Blood creatinine increased (Investigations) | 1
Blood thyroid stimulating hormone increased (Investigations) | 2
Blood urine present (Investigations) | 2
Body temperature increased (Investigations) | 5
Electrocardiogram QT corrected interval prolonged (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Heart rate irregular (Investigations) | 1
Hypoalbuminemia (Investigations) | 1
Hyponatremia (Investigations) | 1
Imaging procedure abnormal (Investigations) | 4
Influenza like illness (Investigations) | 1
Lymphocyte count decreased (Investigations) | 3
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 9
Surgical and medical procedures - Other, specify- Skin biopsy (Investigations) | 1
Weight decreased (Investigations) | 1
Weight gain (Investigations) | 1
Weight increased (Investigations) | 5
Weight loss (Investigations) | 1
Anorexia nervosa (Metabolism and nutrition disorders) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Bartholin's cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Altered state of consciousness (Nervous system disorders) | 1
Confusional state (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Insomnia (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 1
Urinary incontinence (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 1
Micturition urgency (Renal and urinary disorders) | 1
Polyuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Oedema genital (Reproductive system and breast disorders) | 1
Vulvovaginal pain (Reproductive system and breast disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3
Bronchial wall thickening (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders- Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Mucositis management (Surgical and medical procedures) | 1
Embolism (Vascular disorders) | 1
Extremity necrosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 7
Intracranial hemorrhage (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The 5 patients who did not complete the study were for reason other than treatment related toxicities.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-27): https://cdn.clinicaltrials.gov/large-docs/74/NCT02996474/Prot_SAP_000.pdf